CLINICAL TRIAL: NCT02007941
Title: An Open-label, Non-randomized, Parallel-group Design Clinical Trial for Comparative Evaluation of Pharmacokinetics After CKD-501 Between Patients With Renal Impairment and Control Subjects With Normal Renal Function
Brief Title: Comparative Evaluation of Pharmacokinetics After CKD-501 Between Renal Impaired and Normal Renal Function Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19RI113017
Record Dates: First submitted 2013-12-03; First posted 2013-12-11 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Renal Impairment; Healthy
MeSH Terms: conditions — Renal Insufficiency | interventions — lobeglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- End Stage Renal Disease(ESRD) (Experimental): CKD-501 will be administered to patients who have required dialysis and non-dialysis eGFR(estimate glomerular filtration rate ) is Less than 15.
  First, ESRD Patient and normal renal function Subjects are conducted. After the interim analysis, Determine whether early termination or renal impaired subject's progress
  Interventions: Drug: CKD-501
- normal renal function (Active Comparator): CKD-501 will be administered to normal renal function subject who have eGFR(estimate glomerular filtration rate ) of 90 or more.
  First, ESRD Patient and normal renal function Subjects are conducted. After the interim analysis, Determine whether early termination or renal impaired subject's progress
  Interventions: Drug: CKD-501
- Mild renal impairment (Experimental): CKD-501 will be administered to patients who have eGFR(estimate glomerular filtration rate ) is 60 to 89 that.
  Interventions: Drug: CKD-501

INTERVENTIONS:
Drug: CKD-501 — From day 1 to day 3, Once(Day1) CKD-501 0.5mg is administered .
  Other Names: Lobeglitazone

SUMMARY:
The purpose of this study is to assess between the renal impaired patients and normal renal function subjects comparetive evaluation to Pharmacokinetics after CKD-501 Future, When prescription CKD-501 to renal impaired patient, It will be guidelines to provide a basis of instructions.

DETAILED DESCRIPTION:
A Phase 1, Non-randomized, Open, Parallel-Group Clinical trial

ELIGIBILITY:
Inclusion Criteria

All subjects:

* Adult males or females, 20 - 65 years of age (inclusive);
* Body mass index (BMI) range of approximately 18.5-29.9 kg/㎡ (inclusive);
* Agreement with written informed consent
* Agree to Medically acceptable method of contraception during clinical trials

Normal Renal Function subjects:

* Matched to renal impaired patients(ESRD) in the study by age (±7 years), sex and BMI
* Medically healthy with clinically insignificant screening results (e.g., laboratory profiles, medical history, EKG, physical examination);
* eGFR ≥ 90 mL/min/1.73mE2;

Renally impaired subjects:

* Matched to renal impaired patients(ESRD) in the study by age (±7 years), sex and BMI
* Subjects with mild renal impairment (eGFR 60-89 mL/min/1.73mE2) OR moderate renal impairment (eGFR 30-59 mL/min/1.73mE2) OR severe renal impairment (eGFR 15-29 mL/min/1.73mE2) OR dialysis end stage renal disease(ESRD)

Exclusion Criteria

All subjects:

* The subject's systolic blood pressure is outside the range of 100-180mmHg, or diastolic blood pressure is outside the range of 50-110mmHg
* Repeatedly Screening ECG parameters (PR ≥ 210 mse,QRS ≥ 120 msec, QTcF ≥ 500 msec)
* Repeatedly lab(AST >1.25xULN, ALT>1.25xULN ,Total bilirubin >1.5xULN)
* A positive pre-study drug screen.(amphetamines, barbiturates, cocaine, opiates, cannabinoids, benzodiazepin)
* Clinically significant allergic diseases or History of thiazolidinedione class's anaphylaxis reactions
* Can not stop to be taking caffeine (caffeine > 400mg/day), drinking(alcohol > 30 g/day) or severe heavy smoker(cigarette > 10 cigarettes/day) during clinical trials
* Consumption of food which may affect study within 7 days prior to first dose of study medication or taking a dietary supplement now or continued.
* Consumption of drug which may affect study within 7 days prior to first dose of study medication.
* Previously donate whole blood within 60 days or component blood within 30 days prior to first dose of study medication.
* blood transfusion within 30 days prior to first dose of study medication.
* Subjects with participation in another clinical trial within 60 days prior to the study
* An impossible one who participates in clinical trial by Principal investigator's decision

Normal Renal Function subjects:

* Subjects with a history of chronic disease or an acute illness within 28 days of study medication administration
* Subjects with a history of gastrointestinal disease effected study medication or surgery(except appendectomy, hernia surgery)
* Current or chronic history of liver disease or ascites or hepatic encephalopathy

Renally impaired subjects:

* Type I diabetes, Diabetic ketoacidosis, diabetic coma or a history of coma (controllable Type II diabetes including possible)
* Uncontrollable hypertension or severe heart failure
* require treatment with steroid or immunosuppressive drug
* History of renal transplant or undergoing other dialysis method except hemodialysis
* Needs treatment for acute disease, uncontrolled other disease or diabetic complications
* Current or chronic history of liver disease or ascites or hepatic encephalopathy
* Subjects with a history of chronic disease or an acute illness within 28 days of study medication administration
* Subjects with a history of gastrointestinal disease effected study medication or surgery(except appendectomy, hernia surgery)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic( Cmax, AUCt ) of lobeglitazone(CKD-501) Between Renal Impaired patients and Normal Renal function subjects | 0-48 hrs
  * Blood sampling timepoint : (Day 1) 0hr, 0.33hr, 0.66hr, 1hr, 1.5hr, 2hr, 3hr, 6hr, 12hr, 24hr (Day 2)36hr (Day3)48hr- total 12 timepoints per period
  * Additional Blood sampling for unbound fraction analysis : (Day 1) 1hr, 6hr, 12hr
  * Urine collection : (Day 1)0-6hr, 6-12hr, 12-24hr (Day 2) 24-36hr, 36-48hr

SECONDARY OUTCOMES:
The pharmacokinetic( Cmax, AUCt ) of main metabolites(M7) of CKD-501 Between Renal Impaired patients and Normal Renal function subjects | 0-48 hrs
  * Blood sampling timepoint : (Day 1) 0hr, 0.33hr, 0.66hr, 1hr, 1.5hr, 2hr, 3hr, 6hr, 12hr, 24hr (Day 2)12hr (Day3)0hr- total 12 timepoints per period
  * Urine collection : (Day 1)0-6hr, 6-12hr, 12-24hr (Day 2) 24-36hr, 36-48hr

CONTACTS AND LOCATIONS:
Overall Officials: Jae Kuk Shin, Ph.D. M.D, Principal Investigator — The Inje University Busan Paik Hospital
Locations (1):
- The Inje University Busan Paik Hospital, Busan, South Korea